CLINICAL TRIAL: NCT04678869
Title: CiproPAL (Ciprofloxacin Prophylaxis in Acute Leukaemia): A Randomised Trial to Assess the Use of Ciprofloxacin Prophylaxis to Prevent Bacterial Infection in Children Treated on the Induction Phase of the ALLTogether-1 Treatment Protocol
Brief Title: CiproPAL (Ciprofloxacin Prophylaxis in Acute Leukaemia)
Acronym: CiproPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CiproPAL (129038)
Record Dates: First submitted 2020-12-05; First posted 2020-12-22 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Acute Lymphoblastic Leukaemia - Category
Keywords: antibiotic prophylaxis
MeSH Terms: interventions — Ciprofloxacin; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Randomised trial of prophylactic ciprofloxacin (10mg/kg BD, enteral/IV) versus standard of care during the neutropenic period of induction (with an internal pilot study) in patients aged 1-17 years with de-novo ALL treated on ALLTogether-1. Exclusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cirprofloxacin prophylaxis (Experimental): prophylactic ciprofloxacin (10mg/kg BD, enteral/IV)
  Interventions: Drug: Ciprofloxacin
- Standard of care (Active Comparator): standard of care
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Ciprofloxacin — prophylactic ciprofloxacin (10mg/kg BD, enteral/IV)
  Arms: Cirprofloxacin prophylaxis
Drug: Antibiotic — Standard of care antibiotic as per local policy
  Arms: Standard of care

SUMMARY:
CiproPAL is a randomised trial comparing daily ciprofloxacin with local standard care during the induction phase of paediatric ALL treatment, and aims:

1. To assess the efficacy of ciprofloxacin prophylaxis in the reduction of infection during the induction phase of treatment for paediatric Acute Lymphoblastic Leukaemia within the ALLTogether-1 Trial.
2. To evaluate the impact of ciprofloxacin prophylaxis on antimicrobial resistance, both of invasive infections and colonising organisms.

DETAILED DESCRIPTION:
This is a multi-centre randomised trial of prophylactic ciprofloxacin (10mg/kg BD, enteral/IV) versus standard of care during the neutropenic period of induction (with an internal pilot study) in patients aged 1-17 years with de-novo ALL treated on ALLTogether-1. Exclusion criteria include: patients with Down syndrome (who already receive ciprofloxacin prophylaxis), contraindication to fluoroquinolones, non-consent to ALLTogether-1 or CiproPAL. AMR of colonising organisms will be assessed with stool or peri-rectal swab cultures performed at five timepoints within the first year. Longer term invasive infection AMR monitoring will include sensitivity testing of all organisms isolated in confirmed infection for the duration of ALLTogether-1.

The primary outcome is the rate of sterile site bacterial infections during induction, evaluated by intention to treat analysis. Secondary outcomes include rates of febrile episodes, febrile neutropenia, severe infection and infection-related death; rates of AMR; antibiotic exposure; secondary infections; and quinolone side effects. A model-based health economic analysis will be undertaken. Using a conservative effect estimate of 40% reduction in bacteraemia (i.e. a reduction from 15% to 9%) 1052 patients randomised 1:1 gives 85% power with a 5% 2-sided alpha.

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients (1-17 years inclusive) with de-novo Acute Lymphoblastic Leukaemia treated on ALLTogether-1 in the UK in the first 5 days of therapy, up to 14 days is acceptable.
* Written informed consent

Exclusion Criteria:

* Non-participants of the ALLTogether-1 trial
* Patients with Down syndrome who already receive ciprofloxacin prophylaxis
* Chronic active arthritis
* Other contraindication to fluoroquinolones

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1052 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of sterile site bacterial infections during induction | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  rate of sterile site bacterial infections during induction

SECONDARY OUTCOMES:
rates of febrile episodes | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  rates of febrile episodes
rates of febrile neutropenia | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  rates of febrile neutropenia
rates of severe infection and infection-related death | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  severe infection rates and deaths from infection
rates of AMR (antimicrobial resistance) | Until the end of trial approx 10 years (from randomisation until the end of trial declaration in 2031)
  rates of AMR
rates of antibiotic exposure | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  rates of antibiotic exposure
rates of secondary infections | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  rates of secondary infections
quinolone side effects | during induction approx 1 month (from randomisation until the start of consolidation, discontinuing protocol antileukaemic therapy or death post induction)
  quinolone side effects

CONTACTS AND LOCATIONS:
Overall Officials: Robert Phillips, Principal Investigator — University of York
Locations (14):
- United Kingdom (14):
  - Royal Aberdeen Children's Hospital, Aberdeen
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Alder Hey Children's Hospital, Liverpool
  - Great Ormond Street Hospital, London
  - Univeristy College Hospital London, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle
  - Nottingham Children's Hospital, Nottingham
  - John Radcliffe Hospital, Oxford
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Requests for de-identified data should be made in writing to the relevant trials group lead at the CR UK and UCL Cancer Trials Centre (https://www.ctc.ucl.ac.uk/DataSampleSharing.aspx)
Supporting Information: Study Protocol, Analytic Code
Access Criteria: See UCL CTC website
URL: https://www.ctc.ucl.ac.uk/DataSampleSharing.aspx